CLINICAL TRIAL: NCT04765007
Title: Efficacy of Mindfulness Therapy in Orofacial Chronic Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, Daniel Rodríguez Almagro, Physiotherapist, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: mindfulness Ujaen
Record Dates: First submitted 2021-02-02; First posted 2021-02-21 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Mindfulness; Chronic Pain; Orofacial Pain
Keywords: mindfulness; chronic pain; orofacial pain
MeSH Terms: conditions — Chronic Pain; Facial Pain | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness group (Experimental): This arm will be treated with a mindfulness-based stress reduction therapy.
  Interventions: Other: mindfulness-based stress reduction
- Control group (Other): This arm will be treated with a minimal intervention.
  Interventions: Other: Minimal intervention

INTERVENTIONS:
Other: mindfulness-based stress reduction — Eight sessions of two hours and a half, one day per week during eight weeks. In addition, patients will perform a day of intensive silent practice of 6-8 hours of duration.
  The content of each session balances three activities: the presentation of a topic, moments of dialogue and group exploration (using appreciative inquiry) and a Mindfulness practice.
  The sessions will take place in online format, through the google meet application
  Other Names: MBSR
  Arms: Mindfulness group
Other: Minimal intervention — A guided meditation program of eight weeks of duration will be provided to the patients and they will be informed about the procedure and the beneficial effects of the therapy.
  Arms: Control group

SUMMARY:
Psychological impairments have a significant role in management and coping of pain in patients with orofacial pain disorders. The response of this kind of pathologies to topical or systemic medications is not predictable and mindfulness breathing and relaxation techniques could present good results since it help patients to accept their problem and to cope it. In consequence, the present study is aimed to evaluate the efficacy of a mindfulness therapy program in management of chronic orofacial pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed of orofacial chronic pain by a physician.

Exclusion Criteria:

* Pain with oncologic origin
* Severe mental disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-05-04 (Estimated); Primary Completion 2021-05-04 (Estimated); Study Completion 2021-10-07 (Estimated)

PRIMARY OUTCOMES:
orofacial pain intensity | pre-intervention
  mean of orofacial pain in the last seven days evaluated with Numeric Pain Rating Scale (NPRS). A scale from 0 to 10, where 0 is considered as no pain and 10 as the worst pain.
orofacial pain intensity | 8 weeks
  mean of orofacial pain in the last seven days evaluated with Numeric Pain Rating Scale (NPRS). A scale from 0 to 10, where 0 is considered as no pain and 10 as the worst pain
orofacial pain intensity | 5 months
  mean of orofacial pain in the last seven daysevaluated with Numeric Pain Rating Scale (NPRS). A scale from 0 to 10, where 0 is considered as no pain and 10 as the worst pain
Symptoms of temporomandibular disorders | pre-intervention
  Evaluation of the presence or absence of symptoms caused by temporomandibular disorders and their severity evaluated with Fonseca Anamnestic Index (FAI).
Symptoms of temporomandibular disorders | 8 weeks
  Evaluation of the presence or absence of symptoms caused by temporomandibular disorders and their severity evaluated with Fonseca Anamnestic Index (FAI).
Symptoms of temporomandibular disorders | 5 months
  Evaluation of the presence or absence of symptoms caused by temporomandibular disorders and their severity evaluated with Fonseca Anamnestic Index (FAI).
Catastrophization of pain | pre-intervention
  Evaluation of pain catastrophization through Pain Catastrophizing Scale (PCS). The PCS is a 13-item self-report questionnaire. Each item is scored from 0 (not at all) to 4 (always), and scores range from 0 to 52.
Catastrophization of pain | 8 weeks
  Evaluation of pain catastrophization through Pain Catastrophizing Scale (PCS). The PCS is a 13-item self-report questionnaire. Each item is scored from 0 (not at all) to 4 (always), and scores range from 0 to 52.
Catastrophization of pain | 5 months
  Evaluation of pain catastrophization through Pain Catastrophizing Scale (PCS). The PCS is a 13-item self-report questionnaire. Each item is scored from 0 (not at all) to 4 (always), and scores range from 0 to 52.
Kinesiophobia | pre-intervention
  Assessment of fear of movement in temporomandibular disorders evaluated with Tampa Scale of Kinesiophobia for Temporomandibular Disroders (TSK-TMD). The TSK-TMD is an 18-item self-report questionnaire, where the degree of agreement with each of the presented statements is recorded on a response scale from 1 (completely disagree) to 4 (completely agree). The scores are summed to provide a total score, with higher values reflecting greater kinesiophobia.
Kinesiophobia | 8 weeks
  Assessment of fear of movement in temporomandibular disorders evaluated with Tampa Scale of Kinesiophobia for Temporomandibular Disroders (TSK-TMD). The TSK-TMD is an 18-item self-report questionnaire, where the degree of agreement with each of the presented statements is recorded on a response scale from 1 (completely disagree) to 4 (completely agree). The scores are summed to provide a total score, with higher values reflecting greater kinesiophobia.
Kinesiophobia | 5 months
  Assessment of fear of movement in temporomandibular disorders evaluated with Tampa Scale of Kinesiophobia for Temporomandibular Disroders (TSK-TMD). The TSK-TMD is an 18-item self-report questionnaire, where the degree of agreement with each of the presented statements is recorded on a response scale from 1 (completely disagree) to 4 (completely agree). The scores are summed to provide a total score, with higher values reflecting greater kinesiophobia.
Impact of headache | pre-intervention
  Evaluation of the impact caused by headache using the Headache Impact Test (HIT-6)
Impact of headache | 8 weeks
  Evaluation of the impact caused by headache using the Headache Impact Test (HIT-6)
Impact of headache | 5 months
  Evaluation of the impact caused by headache using the Headache Impact Test (HIT-6)
Sleep quality | pre-intervention
  Assessment of sleep quality with the Medical Outcomes Study Sleep Scale (MOS-SS). the MOS-SS is a self-administered questionnaire comprised of 12 items in six different domains or sub-scales.
Sleep quality | 8 weeks
  Assessment of sleep quality with the Medical Outcomes Study Sleep Scale (MOS-SS). the MOS-SS is a self-administered questionnaire comprised of 12 items in six different domains or sub-scales.
Sleep quality | 5 months
  Assessment of sleep quality with the Medical Outcomes Study Sleep Scale (MOS-SS). the MOS-SS is a self-administered questionnaire comprised of 12 items in six different domains or sub-scales.
Dizziness-related disability | pre-intervention
  Evaluation of dizziness-related disability through Dizziness Handicap Inventory (DHI)
Dizziness-related disability | 8 weeks
  Evaluation of dizziness-related disability through Dizziness Handicap Inventory (DHI)
Dizziness-related disability | 5 months
  Evaluation of dizziness-related disability through Dizziness Handicap Inventory (DHI)
Neck pain-related disability | pre-intervention
  Assessment of neck pain-related disability with Neck Disability Index (NDI)
Neck pain-related disability | 8 weeks
  Assessment of neck pain-related disability with Neck Disability Index (NDI)
Neck pain-related disability | 5 months
  Assessment of neck pain-related disability with Neck Disability Index (NDI)